CLINICAL TRIAL: NCT02910596
Title: Effectiveness of Bethanechol Chloride and Early Bladder Training for Prevention of Bladder Dysfunction After Radical Hysterectomy in Cervical Cancer Stage IB - IIA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RJBLA
Record Dates: First submitted 2016-09-20; First posted 2016-09-22 (Estimated); Last update posted 2020-10-23 (Actual); Status verified 2016-09

CONDITIONS: Bladder Dysfunction
MeSH Terms: interventions — Bethanechol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Experimental): * Ucholine(Bethanechol chloride, 10 mg) 2 tablets oral tid, ac Start on 3rd - 5th postoperative day
  * In bethanechol chloride arm arm should be vital signs were monitored every 30 minute on first hour then every 4 hours on first day. Any adverse event were recorded.
  * Remove urethral catheter on 5thpostoperative day. Void volume and postvoid residual urine were record. Intermittent urethral catheterization was used to measure postvoid residual urine. If postvoid residual urine was more than 100 cc in two consecutive measurement, the urethral catheter was reinserted, and medication would be continue until the catheter cloud be removed but medication were not given for more than 1 month. Postvoid residual urine, urinalysis were evaluated at 1 month postoperative
  Interventions: Drug: bethanechol chloride
- B (Experimental): * Early bladder training Start on 3rd - 5th postoperative day
  * Remove urethral catheter on 5th postoperative day. Void volume and postvoid residual urine were recorded. Intermittent urethral catheterization was used to measure postvoid residual urine. If postvoid residual urine was more than 100 cc in two consecutive measurement, the urethral catheter was reinserted, and medication would be continue until the catheter cloud be removed but medication were not given for more than 1 month. Postvoid residual urine, urinalysis were evaluated at 1 month postoperative
  Interventions: Device: early bladder training
- C (Experimental): * Early bladder training and Ucholine(Bethanechol chloride, 10 mg) 2 tablets oral tid, ac Start on 3rd - 5th postoperative day
  * should be vital signs were monitored every 30 minute on first hour then every 4 hours on first day. Any adverse event were recorded.
  * Remove urethral catheter on 5th postoperative day. Void volume and postvoid residual urine were recorded. Intermittent urethral catheterization was used to measure postvoid residual urine. If postvoid residual urine was more than 100 cc in two consecutive measurement, the urethral catheter was reinserted, and medication would be continue until the catheter cloud be removed but medication were not given for more than 1 month. Postvoid residual urine, urinalysis were evaluated at 1 month postoperative
  Interventions: Other: early bladder training and bethanechol chloride
- D (Other): -Remove urethral catheter on 5th postoperative day. Void volume and postvoid residual urine were recorded. Intermittent urethral catheterization was used to measure postvoid residual urine. If postvoid residual urine was more than 100 cc in two consecutive measurement, the urethral catheter was reinserted, and medication would be continue until the catheter cloud be removed but medication were not given for more than 1 month. Postvoid residual urine, urinalysis were evaluated at 1 month postoperative
  Interventions: Other: no early bladder training and no bethanechol chloride

INTERVENTIONS:
Drug: bethanechol chloride — bethanechol chloride(10) 2 tablets oral tid, ac. Start on3rd - 5th postoperative day
  Arms: A
Device: early bladder training — early bladder training start on 3rd - 5thpostoperative day
  Arms: B
Other: early bladder training and bethanechol chloride — bethanechol chloride 2 tablets oral tid, ac and early bladder training start on 3rd - 5th postoperative day
  Arms: C
Other: no early bladder training and no bethanechol chloride — no bethanechol chloride and no early bladder training
  Arms: D

SUMMARY:
Compare the effectiveness of bethanechol chloride and early bladder training for prevention of bladder dysfunction after radical hysterectomy in cervical cancer stage IB - IIA.

DETAILED DESCRIPTION:
Cervical cancer is the third most common cancer in women worldwide, after breast and colorectal cancer. Molecular biology has firmly established a causal relationship between persistent infection with high risk human papilloma virus (HPV) genotypes and cervical cancer.

Cervical cancer stage IB1 and selected IIA 1 lesions without extensive vaginal involvement can be treated with either RH and pelvic lymph node dissection (PLD) or primary chemoradiation.

Bladder dysfunction is the most common complication after radical hysterectomy. The incidence is approximate 10-80 %. Management of bladder dysfunction is continuous urethral catheterization or clean intermittent self-catheterization. Prolonged urethral catheterization may increase the risk of urinary tract infection.

Early postoperative bladder training that consist of a scheduled clamping trans-urethral catheter every 3 h and unclamping trans-urethral catheter 15 min during the entire day.

Bethanechol chloride is a cholinergic drug and may enhance the detrusor muscle contraction, resulting in higher maximum flow rate, and lower postvoid residual urine.

This study was conducted to compare the effectiveness of bethanechol chloride and early bladder training for prevention of bladder dysfunction after radical hysterectomy in cervical cancer stage IB - IIA.

ELIGIBILITY:
Inclusion Criteria:

* Women with cervical cancer stage IB - IIA underwent standard type III radical hysterectomy, both open and laparoscopic approach
* Patient aged 20 - 65 years
* Patient able to give free and informed consent and who agrees to participate be signing the consent form

Exclusion Criteria:

* Patient who had an allergic reaction to bethanechol chloride
* Patient who had neurogenic bladder

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Duration of retrained urethral catheterization(day) after standard type III radical hysterectomy | 5 days postoperative

SECONDARY OUTCOMES:
Rate of urethral catheter removal at 5 days postoperative | 5 days postoperative
Incidence of urinary tract infection at 28 days postoperative | 28 days postoperative
Volume of postvoid residual urine at 28 days postoperative | 28 days postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Narisa Jenrungrojsakul, MD, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No